CLINICAL TRIAL: NCT02315157
Title: Phase I Study of Escalating-Doses of Bendamustine for Patients With Previously Treated Multiple Myeloma
Brief Title: Bendamustine Hydrochloride in Treating Patients With Previously Treated Multiple Myeloma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawn by PI
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14D.244; 2014-009 (Other: CCRRC); JT 5775 (Other: JeffTrial Number)
Record Dates: First submitted 2014-12-09; First posted 2014-12-11 (Estimated); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Multiple Myeloma; Plasma Cell Leukemia
Keywords: Partial Response
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Plasma Cell | interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bendamustine 200 mg/m2 (Experimental): Patients receive bendamustine hydrochloride IV over 60-180 minutes on days 1 and 2 (total dose 400 mg/m2).
  Interventions: Drug: Bendamustine
- Bendamustine 250 mg/m2 (Experimental): Patients receive bendamustine hydrochloride IV over 60-180 minutes on days 1 and 2 (total dose 500 mg/m2).
  Interventions: Drug: Bendamustine

INTERVENTIONS:
Drug: Bendamustine — Given IV
  Other Names: Treakisym; Ribomustin; Levact; Treanda; SDX-105

SUMMARY:
This phase I trial studies the side effects and best dose of bendamustine hydrochloride in treating patients with previously treated multiple myeloma. Drugs used in chemotherapy, such as bendamustine hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify a maximum tolerated dose of bendamustine (bendamustine hydrochloride) in patients with multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the safety of escalating doses of bendamustine in patients with multiple myeloma.

II. To describe the response after bendamustine

OUTLINE: This is a dose-escalation study.

Patients receive bendamustine hydrochloride intravenously (IV) over 60-180 minutes on days 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with multiple myeloma who have not achieved a CR following at least 4 cycles of induction therapy
2. Age up to 80 years
3. ECOG Performance Status of 0 or 1
4. Left ventricular ejection fraction =/> 40%. No uncontrolled arrhythmias or symptomatic cardiac disease
5. FEV1, FVC and DLCO =/> 40%. No symptomatic pulmonary disease.
6. Serum bilirubin <2 x upper limit of normal, alkaline phosphatase <3 x upper limit of normal. No evidence of chronic active hepatitis or cirrhosis. No effusion or ascites > 1 L prior to drainage.
7. HIV negative
8. Negative beta HCG test in woman with child bearing potential, defined as not post-menopausal for 12 months or no previous sterilization
9. Patients or guardian able to sign informed consent
10. Availability of previously collected autologous stem cells (at least 3.0 x 106 CD34 cells/kg)
11. Calculated GFR > 50 ml/minute

Exclusion Criteria:

1. Patients with uncontrolled hypertension (systolic > 140, diastolic > 90 despite antihypertensive therapy
2. Patients with uncontrolled bacteria, viral or fungal infections (currently taking medication and progression of clinical symptoms)
3. New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
4. Relapsed/refractory myeloma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of bendamustine | 2 days
  Defined as the dose where no more than 1 out of 6 patients experience dose-limiting toxicities. Toxicities will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Incidence of toxicity (NCI CTCAE version 4.0) | Up to 92 days following the last administration of study treatment
  Graded according to NCI CTCAE version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Manish Sharma, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Sidney Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Jefferson University Hospitals — http://hospitals.jefferson.edu/